CLINICAL TRIAL: NCT02485457
Title: Validation of NICOM for the Detection of Modification of Stroke Volume
Brief Title: Validation of Nicom Device to Measure Stoke Volume Variation
Acronym: NICOM-VAL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties of recrutment
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2014/17
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Anesthesia
MeSH Terms: interventions — Ringer's Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low volume (Experimental): The protocol will follow the following steps :
  * basal measurements (heart rate, arterial pressure, stroke volume estimated by esophageal Doppler, stoke volume estimated by Nicom)
  * followed by passive leg rising and additional measurements (heart rate, arterial pressure, stoke volume estimated by esophageal Doppler, stoke volume estimated by Nicom)
  * second basal measurements (heart rate, arterial pressure, stoke volume estimated by esophageal Doppler, stoke volume estimated by Nicom)
  * followed by low volume loading (250 ml of Ringer solution) and additional measurements (heart rate, arterial pressure, stoke volume estimated by esophageal Doppler, stoke volume estimated by Nicom)
  Interventions: Procedure: Volume loading; Drug: Ringer solution
- High volume (Experimental): The protocol will follow the following steps :
  * basal measurements (heart rate, arterial pressure, stroke volume estimated by esophageal Doppler, stoke volume estimated by Nicom)
  * followed by passive leg rising and additional measurements (heart rate, arterial pressure, stoke volume estimated by esophageal Doppler, stoke volume estimated by Nicom)
  * second basal measurements (heart rate, arterial pressure, stoke volume estimated by esophageal Doppler, stoke volume estimated by Nicom)
  * followed by low volume loading (500 ml of Ringer solution) and additional measurements (heart rate, arterial pressure, stoke volume estimated by esophageal Doppler, stoke volume estimated by Nicom)
  Interventions: Procedure: Volume loading; Drug: Ringer solution

INTERVENTIONS:
Procedure: Volume loading — Volume loading with Ringer Lactate
Drug: Ringer solution

SUMMARY:
The purpose of this study is to evaluate the ability of NICOM (Noninvasive cardiac output monitor) to detect stroke volume variation induced by leg raising or fluid expansion during surgery

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing general anesthesia with an expected duration exceeding two hours
* gastrointestinal surgery, urological or gynecological surgery.

Exclusion Criteria:

* Difficulty of venous access.
* Contraindication for the use of oesophageal Doppler
* Contraindication for the use of Nicom
* Contraindication for the use of bispectral index
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-06-28 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-12 (Actual)

PRIMARY OUTCOMES:
Stroke volume variation | 6 hours
  Stroke volumes measured by esophageal Doppler and by Nicom: at baseline, after leg passive rising, and after volume loading

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Lariboisière, Paris
  - Marc Fischler, Paris